CLINICAL TRIAL: NCT06275828
Title: The Effect of Perioperative Music Reduces Pain Perception After Anterior Cruciate Ligament Reconstruction.
Brief Title: The Effect of Perioperative and Postoperative Music Reduces Pain Perception After Anterior Cruciate Ligament Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Police General Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Peerapat Tansakul, Director, Police General Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PoliceGeneralHospiral
Record Dates: First submitted 2024-01-27; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: anterior cruciate ligament reconstruction; music therapy; postoperative pain; pain score; anxiety
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- intervention (Experimental)
  Interventions: Device: slow beat mesic listening by headphone

INTERVENTIONS:
Device: slow beat mesic listening by headphone — classic slow beat type from researcher
  Arms: intervention

SUMMARY:
study the effect of music therapy in pre-operative and post operative period and measure the out come by the visual analog scale (pain score) and analgesic drug use such as morphine and the anxiety score

DETAILED DESCRIPTION:
Objectives Primary Objective : To study and compare pain symptoms between the group of patients after undergoing Anterior Cruciate Ligament reconstruction surgery and the control group, using pain relievers along with listening to music perioperatively and postoperatively.

Secondary Objective : To study and compare the levels of anxiety and changes in the circulatory system among patients after undergoing Anterior Cruciate Ligament reconstruction surgery and the control group, from listening to music perioperatively and postoperatively.

Research Questions Does listening to music perioperatively and postoperatively during Arthroscopic Anterior Cruciate Ligament reconstruction surgery help reduce postoperative pain?

Hypothesis The group of patients who listened to music perioperatively and postoperatively during Arthroscopic Anterior Cruciate Ligament reconstruction surgery will experience reduced postoperative pain compared to the group that did not listen to music.

Methodology Randomized Controlled Trial (RCT) Sample Size Calculation The calculation of the sample size for testing two independent means, using the method referenced from the study by Xavier C. Simcock and colleagues on "Intraoperative Music Reduces Perceived Pain After Total Knee Arthroplasty total 38 and add 20% for dropout rate

Inclusion criteria

1. Patient age : More than 18 years old
2. The patient have diagnosis ACL injury by MRI and go on surgery by arthroscopic surgery Exclusion criteria

1. History of knee surgery before this visit 2. ACL injury with multiple ligament injury 3. Hearing loss 4. Denial to surgery or include to study

Study Design & Method This study was a randomized control trial of patient knowns ACL injury and undergoing arthroscopic ACL reconstruction surgery between 2022 to 2023. A total 46 patients were included 23 patients in intervention and 23patients in control group. All patients were evaluated using VAS and anxiety scale preoperative and postoperative and intravenous analgesic drug use at 1,3,12,24,48,72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Anterior cruciate ligament tear from MRI
* Plan to surgery by arthroscopic ACL reconstruction
* must able to listening music from headphone

Exclusion Criteria:

* Hearing problem
* History of morphine and pethidine allergy
* History of previous knee surgery
* intraoperative finding multiple ligament injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | post op 1,3,12,24,48,72 hours before discharge from hospital
  pain score from 0 to 10 (0=no pain, 10=Worst pain)

SECONDARY OUTCOMES:
analgesic drug use | post op 1,3,12,24,48,72 hours before discharge from hospital
  dose of analgesic drug use (morphine, pethidine)
Amsterdam Preoperative Anxiety and Information Scale | pre-operative and post operative at ward
  Score from 6(Least anxiety) to 30(maximum anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Police General Hospital, Bangkok, Pathuwam, Thailand

IPD SHARING:
Plan to Share IPD: No